CLINICAL TRIAL: NCT00002775
Title: PHASE I/II STUDY OF DOCETAXEL (TAXOTERE) AND ESTRAMUSTINE COMBINATION CHEMOTHERAPY IN PATIENTS WITH PROSTATE CANCER
Brief Title: Docetaxel Plus Estramustine in Treating Patients With Metastatic Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064755; CPMC-IRB-7386; NCI-V96-0888
Record Dates: First submitted 1999-11-01; First posted 2004-09-02 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2000-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Estramustine

INTERVENTIONS:
Drug: docetaxel
Drug: estramustine phosphate sodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining docetaxel and estramustine in treating patients who have metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose, toxicity, and pharmacokinetic profile of docetaxel in combination with estramustine in patients with metastatic adenocarcinoma of the prostate. II. Determine the safe dose level of this regimen for Phase II evaluation. III. Determine the efficacy of this regimen with evaluation of objective response rate, duration of response, and time to disease progression in these patients. IV. Determine the duration of survival of these patients on this regimen. V. Evaluate the symptomatic and quality of life effects in these patients.

OUTLINE: This is a dose escalation study (phase I). Patients are stratified into one of two risk groups by number of prior chemotherapy regimens (0-2 vs greater than 2) and occurrence and site(s) of prior radiation. Patients receive oral estramustine three times daily beginning 24 hours prior to docetaxel and continuing for 4 days after infusion. Patients receive docetaxel IV over 1 hour every 21 days. Cohorts of 3-6 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is reached (phase I). The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. A minimum of 6 patients receive treatment at the MTD. Phase II: Patients receive docetaxel IV at the MTD from phase I. Treatment continues in the absence of disease progression or unacceptable toxicity for both phases. Quality of life is assessed. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: Approximately 12-37 patients will be accrued for this study within 13-19 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic adenocarcinoma of the prostate Failure of androgen ablation (orchiectomy or luteinizing hormone releasing hormone, flutamide) -Rise in PSA greater than 50% of nadir confirmed by 2 measurements 1 week apart -Appearance of new soft tissue lesions -Appearance of new lesions on bone scan Measurable or evaluable disease No symptomatic ascites, pleural effusions, or peripheral edema greater than trace No brain or leptomeningeal involvement

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 No history of coagulopathy Hepatic: Bilirubin no greater than upper limit of normal (ULN) SGOT or SGPT no greater than 2.0 times ULN Alkaline phosphatase no greater than 5.0 times ULN Renal: Creatinine no greater than 2.0 times ULN Cardiovascular: No myocardial infarction within past 6 months Pulmonary: No prior pulmonary embolus Neurologic: No prior cerebrovascular accident No symptomatic peripheral neuropathy greater than grade 1 No significant neurologic or psychiatric disorder (psychotic disorder, dementia, or seizure) Other: No other prior malignancy within past 5 years, except: Excised or curatively irradiated nonmelanomatous skin cancer No other serious illness or medical condition No active infection

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy Endocrine therapy: At least 4 weeks since prior hormonal therapy Radiotherapy: At least 4 weeks since prior radiotherapy At least 6 weeks since prior isotope therapy No prior radiotherapy to greater than 30% of bone marrow Surgery: Not specified Other: At least 4 weeks since prior investigational drugs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 1998-02

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P. Petrylak, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center, New York, New York, United States